CLINICAL TRIAL: NCT04999306
Title: Feasibility Study of a Hypnosis Intervention and a Cognitive Behavioral Therapy Intervention to Reduce Fatigue in Patients Undergoing Chemotherapy for Metastatic Colorectal Cancer
Brief Title: Feasibility of 2 Interventions to Reduce Fatigue in Patients With Chemotherapy for Metastatic Colorectal Cancer
Acronym: COLOFIGHT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2021-07 COL; 2021-A01031-40 (Other: ID-RCB)
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer Metastatic
Keywords: hypnosis; Cognitive Behavioral Therapy
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Hypnosis vs Cognitive Behavioral Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental): the sessions will be conducted following the same dynamics and the same exercises (safe place, reification, anchoring): introduction of the session (conversational hypnosis in order to probe the patient's perceptions of his or her illness and fatigue, discussion of myths and realities); induction with the creation of a "safe place" that will be used for each session; visualization; deepening of the trance with work on metaphors (reification technique); making specific suggestions on sensations of fatigue, on regaining energy; then instruction for self-hypnosis or anchoring.
  Interventions: Behavioral: Hypnosis
- CBT group (Experimental): This program will work specifically on the psychosocial determinants of fatigue.
  The first session will be patient education on cancer-related fatigue. S2 will address the concept of perceived control and allow the patient to understand what factors accentuate this condition. S3 will allow the patient to work on the emotions associated with cancer and will be complemented by a hypnosis audio. S4 will address the notion of social support and how the patient can learn to delegate or ask for help. S5 will address the notion of coping strategies, the patient will then be able to identify what he/she puts in place, what is productive and what is not. Finally, the S6 will be a synthesis session that will allow to come back to the points that deserve to be deepened.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: Hypnosis — one weekly session during 6 weeks (6 sessions of 30min/1 hour).
  Arms: Hypnosis group
Behavioral: CBT — one weekly session during 6 weeks (6 sessions of 1 hour).
  Arms: CBT group

SUMMARY:
In patients with colorectal cancer, fatigue ranks as the number one chemotherapy-related adverse event, with 75% of patients experiencing grade 3-4 physical and psychological consequences. Metastatic progression and increasing number of courses of chemotherapy are also aggravating factors.

In this study, the investigator will evaluate the feasibility of two standardized interventions aimed at reducing fatigue in patients with metastatic colorectal cancer. One of the two interventions will focus on hypnosis sessions while the other will implement Cognitive Behavioral Therapy (CBT) sessions.

DETAILED DESCRIPTION:
In patients with cancer, fatigue appears to be one of the most common and persistent symptoms, reported by patients as severe and intense. In a previous observational study, the investigator identified fatigue trajectories of patients undergoing chemotherapy for metastatic colorectal cancer. the investigator were able to show an association between each trajectory and survival curves, where intense fatigue is associated with poor survival rate. Moreover, the investigator were able to identify psychosocial predictors of this fatigue: significant emotional distress, poor adjustment (inadequate coping strategy) and low perceived control over the evolution of the disease. the investigator know that psychosocial intervention programs can act on these variables.

Among the psychosocial interventions, there are Cognitive and Behavioral Therapies (CBT), which are defined as a "new learning that corrects pathological or maladaptive behavior". They are based on an experimental scientific approach and are inspired by behaviorist theories. The effectiveness of CBT in the management of cancer-related symptoms, including sleep problems and fatigue, has been demonstrated by several authors. However, these therapies are too often implemented in non-standardized studies (no specific protocol, little evaluation, and difficult replication), or are confounded with other complementary therapies.

In order to improve the management of fatigue, hypnosis also seems to be an interesting approach. The French National Academy of Medicine, in its report on complementary therapies of March 2013, underlines the interest of hypnosis in the management of the chemotherapy side effects. Studies in breast cancer patients show a positive effect of hypnosis combined with CBT on symptoms of distress and physical fatigue. However, like CBT, there is a lack of standardized studies on the subject.

Therefore, before conducting a Randomized Controlled Trial (RCT), a feasibility study seems essential to measure the proportion of volunteers who want to participate in this study as well as the acceptability of the program and the method of data collection.

In this study, the investigator will evaluate the feasibility of two standardized interventions (hypnosis and CBT) aimed at reducing fatigue in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* World Health Organization (WHO) status ≤ 2
* Colorectal adenocarcinoma in progression after first line metastatic chemotherapy
* Able to understand and read French
* Visual Analog Scale (VAS) fatigue ≥ 4
* Patient starting a second or third line of metastatic chemotherapy
* Patient having signed the informed consent
* Patient subscribing to a French Social Security system

Exclusion Criteria:

* Patients without phones or devices for sessions at home
* Bradycardia (< 50 beats/minute) with β-blockers
* Known severe heart failure with ventricular ejection fraction < 40%.
* Presence of known or symptomatic brain metastases
* Chronic pain evolving for more than three months and using morphine
* Patient used to and having a regular and habitual practice of relaxation techniques such as yoga, hypnosis, sophrology, meditation.
* Medical (neurological, psychiatric, etc.) or psychological conditions that do not allow participation in the protocol (filling out the questionnaires, the booklet, as well as following the sessions)
* Hearing-impaired patient without hearing aids
* Patient under guardianship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
patient adherent to the program. | From first session to sixth session
  Proportion of patient adherent to the program: A patient will be considered adherent if he/she participates in at least 4 of the 6 intervention sessions.

SECONDARY OUTCOMES:
acceptance of participation in the study | At the inclusion
  Proportion of patients giving their consent to participate in the study relative to patients to whom the study was proposed
reasons for non-adherence to the program | At 2 weeks post intervention
  Individual semi-directive interview to understand the non-adherence to the program
To highlight the barriers/facilitators to the implementation of the protocol | At 2 weeks post intervention
  Individual semi-directive interview to assessed the Barriers/facilitators to the implementation of the protocol
Client Satisfaction Questionnaire-Core 8 (CSQ-8) | At 2 weeks post intervention
  Self-report statement of satisfaction with health and human services. The CSQ-8 contains 8 items organized into 4-point Likert. For overall score, sum item responses, range from 8-32, higher score indicates higher satisfaction.
Visual Analog Scale of Fatigue | At inclusion, daily during all the intervention to 2 weeks post intervention, at 3 months post-intervention
  Numeric rating scales 0 (no fatigue) to 10 (maximum fatigue)
Multidimensional Fatigue Inventory-Core 20 (MFI20) | At inclusion, at 2 weeks post intervention and at 3 months post-intervention
  The Multidimensional Fatigue Inventory (MFI-20) developed basically to assess 5 main kinds of fatigue: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity.
  The MFI20 contains 20 items that measure the previously mentioned dimension of fatigue. Each item ask the individuals to mark on a (1-5 or 1-7) point rating scale to what extent the statement "is true" and applies to them or "not true".
Quality of life questionnaire-Core 30 (QLQ-C30) | At inclusion, at 2 weeks post intervention and at 3 months post-intervention
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Portales, MD, Study Chair — Montpellier Cancer Institut (ICM); Louise Baussard, PhD, Study Chair — University of Nimes
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone P, Richardson A, Ream E, Smith AG, Kerr DJ, Kearney N. Cancer-related fatigue: inevitable, unimportant and untreatable? Results of a multi-centre patient survey. Cancer Fatigue Forum. Ann Oncol. 2000 Aug;11(8):971-5. doi: 10.1023/a:1008318932641. PMID 11038033
- [Background] Forlenza MJ, Hall P, Lichtenstein P, Evengard B, Sullivan PF. Epidemiology of cancer-related fatigue in the Swedish twin registry. Cancer. 2005 Nov 1;104(9):2022-31. doi: 10.1002/cncr.21373. PMID 16206253
- [Background] Lawrence DP, Kupelnick B, Miller K, Devine D, Lau J. Evidence report on the occurrence, assessment, and treatment of fatigue in cancer patients. J Natl Cancer Inst Monogr. 2004;(32):40-50. doi: 10.1093/jncimonographs/lgh027. PMID 15263040
- [Background] Kangas M, Bovbjerg DH, Montgomery GH. Cancer-related fatigue: a systematic and meta-analytic review of non-pharmacological therapies for cancer patients. Psychol Bull. 2008 Sep;134(5):700-741. doi: 10.1037/a0012825. PMID 18729569
- [Background] Mustian KM, Alfano CM, Heckler C, Kleckner AS, Kleckner IR, Leach CR, Mohr D, Palesh OG, Peppone LJ, Piper BF, Scarpato J, Smith T, Sprod LK, Miller SM. Comparison of Pharmaceutical, Psychological, and Exercise Treatments for Cancer-Related Fatigue: A Meta-analysis. JAMA Oncol. 2017 Jul 1;3(7):961-968. doi: 10.1001/jamaoncol.2016.6914. PMID 28253393
- [Background] Berger AM, Kuhn BR, Farr LA, Lynch JC, Agrawal S, Chamberlain J, Von Essen SG. Behavioral therapy intervention trial to improve sleep quality and cancer-related fatigue. Psychooncology. 2009 Jun;18(6):634-46. doi: 10.1002/pon.1438. PMID 19090531
- [Background] Cousson-Gelie F, Bruchon-Schweitzer M, Atzeni T, Houede N. Evaluation of a psychosocial intervention on social support, perceived control, coping strategies, emotional distress, and quality of life of breast cancer patients. Psychol Rep. 2011 Jun;108(3):923-42. doi: 10.2466/02.07.15.20.PR0.108.3.923-942. PMID 21879639
- [Background] Page MS, Berger AM, Johnson LB. Putting evidence into practice: evidence-based interventions for sleep-wake disturbances. Clin J Oncol Nurs. 2006 Dec;10(6):753-67. doi: 10.1188/06.CJON.753-767. PMID 17193942
- [Background] Morin CM, Vallieres A, Guay B, Ivers H, Savard J, Merette C, Bastien C, Baillargeon L. Cognitive behavioral therapy, singly and combined with medication, for persistent insomnia: a randomized controlled trial. JAMA. 2009 May 20;301(19):2005-15. doi: 10.1001/jama.2009.682. PMID 19454639
- [Background] Carlson LE, Zelinski E, Toivonen K, Flynn M, Qureshi M, Piedalue KA, Grant R. Mind-Body Therapies in Cancer: What Is the Latest Evidence? Curr Oncol Rep. 2017 Aug 18;19(10):67. doi: 10.1007/s11912-017-0626-1. PMID 28822063
- [Background] Barsevick AM, Irwin MR, Hinds P, Miller A, Berger A, Jacobsen P, Ancoli-Israel S, Reeve BB, Mustian K, O'Mara A, Lai JS, Fisch M, Cella D; National Cancer Institute Clinical Trials Planning Meeting. Recommendations for high-priority research on cancer-related fatigue in children and adults. J Natl Cancer Inst. 2013 Oct 2;105(19):1432-40. doi: 10.1093/jnci/djt242. Epub 2013 Sep 18. PMID 24047960
- [Background] Sood A, Barton DL, Bauer BA, Loprinzi CL. A critical review of complementary therapies for cancer-related fatigue. Integr Cancer Ther. 2007 Mar;6(1):8-13. doi: 10.1177/1534735406298143. PMID 17351022
- [Background] Cramer H, Lauche R, Paul A, Langhorst J, Kummel S, Dobos GJ. Hypnosis in breast cancer care: a systematic review of randomized controlled trials. Integr Cancer Ther. 2015 Jan;14(1):5-15. doi: 10.1177/1534735414550035. Epub 2014 Sep 18. PMID 25233905
- [Background] Montgomery GH, Bovbjerg DH, Schnur JB, David D, Goldfarb A, Weltz CR, Schechter C, Graff-Zivin J, Tatrow K, Price DD, Silverstein JH. A randomized clinical trial of a brief hypnosis intervention to control side effects in breast surgery patients. J Natl Cancer Inst. 2007 Sep 5;99(17):1304-12. doi: 10.1093/jnci/djm106. Epub 2007 Aug 28. PMID 17728216
- [Background] Montgomery GH, Sucala M, Baum T, Schnur JB. Hypnosis for Symptom Control in Cancer Patients at the End-of-Life: A Systematic Review. Int J Clin Exp Hypn. 2017 Jul-Sep;65(3):296-307. doi: 10.1080/00207144.2017.1314728. PMID 28506144
- [Background] Jensen MP, Gralow JR, Braden A, Gertz KJ, Fann JR, Syrjala KL. Hypnosis for symptom management in women with breast cancer: a pilot study. Int J Clin Exp Hypn. 2012;60(2):135-59. doi: 10.1080/00207144.2012.648057. PMID 22443523
- [Background] Gentile S, Delaroziere JC, Favre F, Sambuc R, San Marco JL. Validation of the French 'multidimensional fatigue inventory' (MFI 20). Eur J Cancer Care (Engl). 2003 Mar;12(1):58-64. doi: 10.1046/j.1365-2354.2003.00295.x. PMID 12641557
- [Background] Hinz A, Fleischer M, Brahler E, Wirtz H, Bosse-Henck A. Fatigue in patients with sarcoidosis, compared with the general population. Gen Hosp Psychiatry. 2011 Sep-Oct;33(5):462-8. doi: 10.1016/j.genhosppsych.2011.05.009. Epub 2011 Jun 24. PMID 21749844
- [Background] Kuhnt S, Ernst J, Singer S, Ruffer JU, Kortmann RD, Stolzenburg JU, Schwarz R. Fatigue in cancer survivors--prevalence and correlates. Onkologie. 2009 Jun;32(6):312-7. doi: 10.1159/000215943. Epub 2009 May 12. PMID 19521117
- [Background] Singer S, Kuhnt S, Zwerenz R, Eckert K, Hofmeister D, Dietz A, Giesinger J, Hauss J, Papsdorf K, Briest S, Brown A. Age- and sex-standardised prevalence rates of fatigue in a large hospital-based sample of cancer patients. Br J Cancer. 2011 Jul 26;105(3):445-51. doi: 10.1038/bjc.2011.251. Epub 2011 Jul 12. PMID 21750551
- [Background] Askay SW, Patterson DR, Sharar SR. VIRTUAL REALITY HYPNOSIS. Contemp Hypn. 2009 Mar;26(1):40-47. doi: 10.1002/ch.371. PMID 20737029
- [Background] Montgomery GH, David D, Winkel G, Silverstein JH, Bovbjerg DH. The effectiveness of adjunctive hypnosis with surgical patients: a meta-analysis. Anesth Analg. 2002 Jun;94(6):1639-45, table of contents. doi: 10.1097/00000539-200206000-00052. PMID 12032044
- [Background] Schnur JB, Kafer I, Marcus C, Montgomery GH. HYPNOSIS TO MANAGE DISTRESS RELATED TO MEDICAL PROCEDURES: A META-ANALYSIS. Contemp Hypn. 2008 Aug 21;25(3-4):114-128. doi: 10.1002/ch.364. PMID 19746190
- [Background] Montgomery GH, Schnur JB, Kravits K. Hypnosis for cancer care: over 200 years young. CA Cancer J Clin. 2013 Jan;63(1):31-44. doi: 10.3322/caac.21165. Epub 2012 Nov 20. PMID 23168491
- [Background] Gielissen MF, Verhagen S, Witjes F, Bleijenberg G. Effects of cognitive behavior therapy in severely fatigued disease-free cancer patients compared with patients waiting for cognitive behavior therapy: a randomized controlled trial. J Clin Oncol. 2006 Oct 20;24(30):4882-7. doi: 10.1200/JCO.2006.06.8270. PMID 17050873
- [Background] Gielissen MF, Verhagen CA, Bleijenberg G. Cognitive behaviour therapy for fatigued cancer survivors: long-term follow-up. Br J Cancer. 2007 Sep 3;97(5):612-8. doi: 10.1038/sj.bjc.6603899. Epub 2007 Jul 24. PMID 17653075
- [Background] Poort H, Verhagen CA, Peters ME, Goedendorp MM, Donders AR, Hopman MT, Nijhuis-van der Sanden MW, Berends T, Bleijenberg G, Knoop H. Study protocol of the TIRED study: a randomised controlled trial comparing either graded exercise therapy for severe fatigue or cognitive behaviour therapy with usual care in patients with incurable cancer. BMC Cancer. 2017 Jan 28;17(1):81. doi: 10.1186/s12885-017-3076-0. PMID 28129746
- [Derived] Baussard L, Cousson-Gelie F, Jarlier M, Charbonnier E, Le Vigouroux S, Montalescot L, Janiszewski C, Fourchon M, Coutant L, Guerdoux E, Portales F. Hypnosis and cognitive behavioral therapy with online sessions to reduce fatigue in patients undergoing chemotherapy for a metastatic colorectal cancer: Rational and study protocol for a feasibility study. Front Psychol. 2022 Jul 27;13:953711. doi: 10.3389/fpsyg.2022.953711. eCollection 2022. PMID 35967617
- See also: Institut National du Cancer Inc. Les cancers en France — https://www.e-cancer.fr/ressources/cancers_en_france/
- See also: Bontoux D, Couturier D, Menkes C-J. Thérapies complémentaires - acupuncture, hypnose, ostéopathie, tai-chi - leur place parmi les ressources de soins - Académie nationale de médecine | Une institution dans son temps — http://www.academie-medecine.fr/therapies-complementaires-acupuncture-hypnose-osteopathie-tai-chi-leur-place-parmi-les-ressources-de-soins/